CLINICAL TRIAL: NCT03450226
Title: Effects of Stellate Ganglion Block on Hemodynamics Instability During Beating Heart Surgery
Brief Title: Stellate Ganglion Block in Beating Heart Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, sara abdallah, doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SGB in beating heart surgery
Record Dates: First submitted 2018-02-19; First posted 2018-03-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Cardiac Arrythmias
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment (Experimental): patients will receive a stellate ganglion block with 10 ml of 0.25 % bupivacaine
  Interventions: Drug: stellate ganglion block
- control (No Intervention): patients will be controlled

INTERVENTIONS:
Drug: stellate ganglion block — After induction of general anesthesia, patients will receive a stellate ganglion block using a standard and well described paratracheal technique, The patient's head will be extended and a 4-5-cm, 22-gauge needle inserted at the medial edge of the sternocleidomastoid muscle just below the level of the cricoid cartilage at the level of the transverse process of C6 or C7. After advancing to the transverse process the needle will be withdrawn 2-3 mm prior to injection. A negative aspiration test will be performed in two planes before a 1-ml test dose is used to exclude unintentional intravascular injection (vertebral or subclavian arteries) or subarachnoid injection into the dural sleeve.4 A total of 10 ml of 0.25% bupivacaine will be injected.
  Other Names: bupivacaine; marcaine
  Arms: treatment

SUMMARY:
studies suggest that off-pump coronary artery bypass surgery is associated with improved outcomes when compared to on-pump coronary artery bypass. many studies have shown that off-pump coronary bypass surgery reduces patient morbidity and mortality.

manipulation of the coronary arteries during cardiac surgery can stimulate the adjacent post-ganglionic sympathetic fibers and mimic stellate ganglion stimulation ,stellate ganglion block (SGB) can interrupt this reflex by decreasing the efferent cervical sympathetic outflows.

DETAILED DESCRIPTION:
when adopting off-pump surgery , the cardiac surgery team must adopt new techniques to handle a beating heart and the variations in hemodynamics that can occur when performing this type of procedure the incidence rate of cardiac arrhythmia occurring during and after surgery is one of the major complication in open heart surgery. in addition , intraoperative hemodynamic disorders, caused by changes in plasma levels of epinephrine and norepinephrine after surgical stimulation , are some of challenges for patients undergoing off-pump coronary artery bypass surgery. hemodynamic disruption leads to myocardial ischemia, resulting in increased incidence of cardiovascular events and mortality.

stellate ganglion is formed by the fusion of inferior cervical and first thoracic sympathetic ganglia and is located behind the subclavian artery and anterior to the first rib. the inferior cervical cardiac nerves arise from the medial aspect of the stellate ganglia and provide the cardio-accelerator nerve fibers to the cardiac plexus. stellate ganglion stimulation augments peak systolic pressure, and the enhanced myocardial contractility is secondary to stimulation by postganglionic nerve fibers which traverse from stellate ganglion down the great vessels and along the coronary arteries into the myocardium.the blockage of inferior cervical cardiac nerves is responsible for the bradycardia seen following SGB. SGB has been shown to prevent and control perioperative hypertension induced by increased sympathetic activity.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective off-pump coronary artery bypass grafting surgery
* patients with an ejection fraction of more than 50%
* creatinine level of less than 2.0 mg / 100 ml
* no evidence of heart failure
* no significant chronic obstructive lung disease
* age of less than 60 years

Exclusion Criteria:

* emergency surgery
* patients on thrombolytic therapy
* patients with coagulation disorders
* patients requiring heart lung machine
* patients with clinical contraindications to SGB ( including allergy to local anesthetic , carotid vascular disease as defined by ipsilateral prior carotid endarterectomy or carotid stent, superficial infection at the proposed puncture site, contralateral phrenic or laryngeal nerve palsies , and severe chronic obstructive pulmonary disease )
* patients with history of atrial fibrillation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
postoperative electrocardiogram changes | up to 7 days
  absence of new onset postoperative cardiac arrhythmia and myocardial infarction after off-pump coronary artery bypass surgery